CLINICAL TRIAL: NCT03135912
Title: Three-Arm Trial of Novel Treatment for Tinea Pedis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: South End Skin Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SESK-001
Record Dates: First submitted 2016-12-20; First posted 2017-05-02 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Tinea Pedis
Keywords: Tinea Pedis; Athlete's Foot
MeSH Terms: conditions — Tinea Pedis | interventions — Terbinafine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental Treatment (Experimental): Patients supplied with Experimental Drug SESC 01 for daily topical therapy for 4 weeks.
  Interventions: Drug: Experimental Drug SESC 01
- Vehicle Control (Placebo Comparator): Patients supplied with inactive vehicle (placebo), identical to experimental treatment but without active ingredients, to be applied daily for 4 weeks.
  Interventions: Drug: Placebo
- Active Comparator (Active Comparator): Terbinafine hydrochloride cream, to be applied twice daily for 4 weeks.
  Interventions: Drug: Terbinafine Hydrochloride

INTERVENTIONS:
Drug: Experimental Drug SESC 01 — Topical experimental treatment comprising a combination of approved topical therapies and a new dosage method.
  Arms: Experimental Treatment
Drug: Placebo — Dosage method of SESC 01, without active ingredients.
  Arms: Vehicle Control
Drug: Terbinafine Hydrochloride — Topical terbinafine hydrochloride cream.
  Other Names: Lamisil AT
  Arms: Active Comparator

SUMMARY:
This is a three-arm randomized controlled trial to assess the efficacy of an experimental treatment in the treatment of tinea pedis (athlete's foot). The experimental treatment will be tested against a vehicle control to determine efficacy and safety, and against an active comparator to evaluate the success of the treatment relative to an existing gold-standard treatment. Patients will be treated for four weeks, with their condition being assessed at the end of treatment and two weeks after the end of treatment. The primary endpoint for this study is effective treatment rate at the week 6 evaluation, defined as a mycological cure and minimal clinical signs & symptoms. Secondary endpoints include safety and patient evaluation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* male or female, aged 18 or above
* clinical diagnosis of tinea pedis
* diagnosis confirmed with potassium hydroxide microscopy
* availability for the duration of the study (6 weeks)
* willingness to comply with study protocol
* informed consent

Exclusion Criteria:

* moccasin-type tinea pedis
* severe maceration of interdigital spaces
* severe fissuring
* history of dry feet, cracking, fissuring
* concurrent onychomycosis
* serous exudate or pus
* topical antifungal treatment in the past 2 weeks
* systemic antifungal treatment in the past 4 weeks
* concurrent immunosuppressive or antimicrobial therapy
* liver disease
* pregnancy or breastfeeding
* known hypersensitivity to any ingredients of trial agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2017-08-02 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
Effective Treatment (Mycological Cure and Minimal Symptoms) | 6 weeks
  Binary outcome measure defined as mycological cure AND a total clinical assessment score less than or equal to 2 (out of a possible 18). Mycological cure is defined as negative potassium hydroxide microscopy, while the clinical assessment is based on a sum of 6 symptoms (desquamation, vesiculation, erythema, fissuring, maceration, and pruritus) scored 0-3 by a physician.

SECONDARY OUTCOMES:
Rate of Adverse Events | 6 weeks
  To examine treatment safety, we will calculate the rate of adverse events and serious adverse and compare them between the study's three arms using Chi-square tests to evaluate whether a statistically significant difference is present.
Effective Treatment (Mycological Cure and Minimal Symptoms) | 4 weeks
  Effective treatment as defined above, but measured at the end of treatment (4 weeks after the beginning of participation).
Patient Satisfaction Score | 4 weeks
  At the conclusion of treatment, patients complete a brief survey on their impressions of the treatment's tolerability, effectiveness, and convenience on a five-point scale, where 1 = poor, 2 = fair, 3 = good, 4 = very good, 5 = excellent, or they may answer with "No answer/prefer not to say". Scores will be compared for each of the three characteristics and as a sum of the three scores.
Self-Reported Patient Compliance | 4 weeks
  On the same experience questionnaire, patients are asked to estimate how many doses of treatment they missed or forgot to take. Possible answers are None, 1-2, 3-4, 5-6, 7-8, or 9 or more. This indicates whether there is a significant difference in patients' likelihood to adhere to a treatment regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Schanbacher, MD, Principal Investigator — South End Skin Care
Locations (1):
- Kuchnir Dermatology & Dermatologic Surgery, Milford, Massachusetts, United States